CLINICAL TRIAL: NCT00262951
Title: A Phase II Pilot Study of Multi-Agent Neo-Adjuvant Chemoradiation in Patients With Locally Advanced Pancreatic Adenocarcinoma
Brief Title: Chemoradiation in Locally Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed at a planned interim analysis by meeting a predefined toxicity endpoint
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004LS060; 0410M64346 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Results first posted 2012-02-03 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Interferon-alpha; Introns; Cisplatin; Fluorouracil; Radiotherapy; Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pancreatic Adenocarcinoma Patients (Experimental): Pancreatic Adenocarcinoma Patients treated with chemotherapy regimen and radiation (and or surgery).
  Interventions: Biological: recombinant interferon alfa; Drug: cisplatin; Drug: fluorouracil; Radiation: radiation therapy; Procedure: Resection of tumor

INTERVENTIONS:
Biological: recombinant interferon alfa — administered subcutaneously (SQ)at a dose of 3 million units Day 1,3, and 5 each week in Cycle 1
  Other Names: IFN alpha; IFN-alpha-2b
Drug: cisplatin — administered at a dose of 30 mg/m2 intravenously (IV) day 1 each week in Cycle 1
  Other Names: cisplatinum; cis-diamminedichloroplatinum(II) (CDDP)
Drug: fluorouracil — administered at a dose of 175 mg/m^2/day continuous infusion (CI) for 38 days in Cycle 1 and then 500 mg/m^2 intravenously (IV) each week for 6 weeks followed by a 2 week rest (1 cycle = 8 weeks)in Cycle 2 and 3
  Other Names: 5-FU
Radiation: radiation therapy — 5040 cGy total, in 28 fractions, at 180 cGy/fraction daily, Monday -Friday, for 5½ weeks (days 1-5, 8-12, 15-19, 22-26, 29-33, 36-38).
Procedure: Resection of tumor — After Cycle 1 treatment (if resectable)- In the absence of metastatic disease, special emphasis will be paid to the local tumor. Evaluation of the growth/regression of the tumor will be made as it relates to resectability. Surgical exploration will start with a diagnostic laparoscopy. If no evidence of carcinomatosis, liver metastases or other evidence of metastatic disease is encountered, then a laparotomy will be performed. In the absence of clear technical unresectability, a radical pancreaticoduodenectomy, distal or total pancreatectomy (and resection of any involved structures) will be performed as mandated by tumor anatomy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells. Interferon alfa may interfere with the growth of tumor cells. Giving combination chemotherapy and radiation therapy together with interferon alfa before surgery may shrink the tumor so it can be removed. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy and radiation therapy together with interferon alfa works in treating patients with locally advanced pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effect of neoadjuvant chemoradiotherapy and interferon alfa on converting patients with locally advanced unresectable adenocarcinoma of the pancreas to resectability.

Secondary

* Determine the rate and severity of early and late toxic effects of these regimens in these patients.
* Improve surgical morbidity profile and overall survival of patients who undergo surgical resection.
* Determine overall and progression-free survival of patients treated with this regimen.

OUTLINE: This is an pilot, single center study.

* Part 1 (neoadjuvant therapy): Patients receive fluorouracil IV continuously over 24 hours on days 1-38; cisplatin IV over 1 hour on days 1, 8, 15, 22, 29, and 36; and interferon alfa subcutaneously on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, 33, 36, and 38. Patients also undergo radiotherapy on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-38. Patients then undergo restaging. Patients with resectable disease undergo surgery, and 4-10 weeks later, proceed to part 2. Patients with unresectable disease proceed directly to part 2, 4 weeks after completion of neoadjuvant therapy.
* Part 2 (chemotherapy): Patients receive fluorouracil IV on days 1, 8, 15, 22, 29, and 36. Treatment repeats every 56 days for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients with unresectable disease undergo restaging after each course of fluorouracil. If the tumor subsequently becomes resectable, patients then undergo surgery.

After completion of study treatment, patients are followed periodically for 5 years and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have newly diagnosed computated tomography (CT) and endoscopic ultrasound(EUS) stage Tx-4, N0-1, M0 adenocarcinoma of pancreas according to the American Joint Committee on Cancer (AJCC) staging system. The following cell types will NOT be eligible: adenosquamous carcinoma, ampullary carcinoma, carcinoid tumor, cystadenocarcinoma, cystadenoma, distal common bile duct carcinoma, duodenal carcinoma, or islet cell carcinoma
* Treatment must begin within 60 days of diagnosis
* Must have locally advanced inoperable pancreatic cancer with no metastatic spread as determined by a baseline diagnostic CT scan of the chest, endoscopic ultrasound and CT scan with intravenous (IV) contrast (or MRI) of abdomen/pelvis, within 30 days prior to registration.
* No prior systemic chemotherapy or radiation therapy for pancreatic cancer
* Documented Eastern Cooperative Oncology Group (ECOG/Zubrod) performance status 0-1 within 14 days prior to registration
* Adequate hematologic, renal and hepatic function as defined by the following laboratory values (completed within 14 days prior to registration)

  * white blood cell (WBC) > 3,000 mm3
  * absolute neutrophil count (ANC) > 1,500 mm3
  * platelet count ≥ 100,000 mm3
  * hemoglobin > 9.5 g/dl
  * serum creatinine < 1.5 times institutional upper limit of normal (ULN)
  * total bilirubin ≤ 3 mg/dl
  * AST (SGOT) < 4.0 times institutional ULN
  * ALT (SGPT) < 4.0 times institutional ULN
  * alkaline phosphatase < 2.0 times institutional ULN
* Age ≥ 18 years
* Life expectancy ≥ 12 weeks
* Patient (male or female) of reproductive potential are required to use a medically acceptable contraception during treatment and for 3 months after the last dose of chemotherapy.
* Not pregnant or breastfeeding since the drugs used in this study are Pregnancy Category D: Clear evidence of risk in pregnancy. A negative pregnancy test is required within 7 days of registration if pre- or perimenopausal (i.e., last menstrual period within one year of registration)
* If patient has a previous diagnosis of cancer, all of the following criteria must be met and documented in the patient's medical record:

  * Patient has undergone potentially curative therapy for all prior malignancies.
  * No evidence of prior malignancies for at least 5 years (except for successfully treated cervical carcinoma in situ, carcinoma in situ of the breast, or nonmelanoma skin cancer.
  * No evidence of recurrence of any prior malignancy.
* Patient who is receiving chronic immunotherapy (e.g. prednisone or methotrexate) for collagen vascular disease or other chronic immunologic abnormality are not eligible.
* Not requiring one or more of the contraindicated medications
* Patient must be able to understand the potential risks and benefits associated with this study. Patient able to give informed consent and would likely to comply with the study parameters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-01; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward W. Greeno, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients participated in Part 1 of the study only.
Groups:
- Pancreatic Adenocarcinoma Patients: Pancreatic Adenocarcinoma Patients treated with chemotherapy regimen and radiation (and or surgery). Patients were given one cycle of continuous infusion 5-FU (175 mg/m^2/day for 38 days), weekly cisplatin 30 mg/m^2 over 1 hour, and IFN-alpha-2b (3 million units given subcutaneously on days 1, 3, and 5 of each week for 5½ weeks) with radiation therapy (5040 cGy total, in 28 fractions, at 180 cGy/fraction daily, Monday -Friday, for 5½ weeks) followed by two cycles of bolus 5-FU alone (500 mg/m^2 weekly * 6, followed by 2 weeks of rest).
Period: Overall Study
Arm/Group | Pancreatic Adenocarcinoma Patients
Started | 23
Completed | 7
Not Completed | 16
Not completed — Progressive disease/relapse | 3
Not completed — Adverse Event | 7
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Alternative treatment | 3
Not completed — Off treatment for other disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pancreatic Adenocarcinoma Patients
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Whom Tumor Was Resectable
Description: Tumor response is measured in terms of resectability, as measured by CT scan at 2 weeks after completion of each course. A CT scan of the chest abdomen and pelvis will be performed in order to evaluate for the presence of metastatic disease. If no metastatic disease, emphasis will be paid to the local tumor. Evaluation of the growth/regression of the tumor will be made as it relates to resectability. If potential for resection then surgery will be recommended. This protocol will be followed after each cycle.
Time Frame: Up to 5 Years or Until Disease Progression
Measure: Number; unit: Participants
Groups:
- Pancreatic Adenocarcinoma Patients: Pancreatic Adenocarcinoma Patients treated with chemotherapy regimen and radiation (and or surgery). Patients will be given one cycle of continuous infusion 5-FU (175 mg/m^2/day for 38 days), weekly cisplatin 30 mg/m^2 over 1 hour, and IFN-alpha-2b (3 million units given subcutaneously on days 1, 3, and 5 of each week for 5½ weeks) with radiation therapy (5040 cGy total, in 28 fractions, at 180 cGy/fraction daily, Monday -Friday, for 5½ weeks) followed by two cycles of bolus 5-FU alone (500 mg/m^2 weekly * 6, followed by 2 weeks of rest).
Arm/Group | Pancreatic Adenocarcinoma Patients
Number analyzed (Participants) | 23
Participants | 7

2. Secondary Outcome: Overall Survival
Description: In all patients, measured from the date of the patient's registration in this study, until the date of the patient's death or date last known alive (if observation was censored).
Time Frame: Up to 5 Years or Date of Death, Whichever Occurred First
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pancreatic Adenocarcinoma Patients
Number analyzed (Participants) | 23
Months | 11.5 [7.5 to 15.2]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed during study treatment and for 1 month following study treatment (for up to 10 months).
Arm/Group | Pancreatic Adenocarcinoma Patients
Serious Adverse Events (participants affected / at risk) | 12/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pancreatic Adenocarcinoma Patients (N=23)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (2)
Fever (in the absence of neutropenia) (General disorders) | 2 (3)
Weight loss (General disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastritis (including bile reflux) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal, other (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Gallbladder perforation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Melana/Gastrointestinal bleeding (Blood and lymphatic system disorders) | 1 (1)
Upper Gastrointestinal hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Genitourinary hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, other (Blood and lymphatic system disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 1 (1)
Infection with normal absolute neutrophils (Infections and infestations) | 1 (2)
Syncope (fainting) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pain, other (General disorders) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal/genitourinary, other (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pancreatic Adenocarcinoma Patients (N=23)
Blood/Bone Marrow/Other (Blood and lymphatic system disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 11 (16)
Leucocytes/total white blood count (Blood and lymphatic system disorders) | 21 (99)
Neutrophils/granulocytes/absolute neutrophils/absolute granulocyte count (Blood and lymphatic system disorders) | 18 (58)
Platelets (Blood and lymphatic system disorders) | 14 (32)
Fatigue/asthenia/lethargy/malaise (General disorders) | 22 (46)
Fever in the absence of neutropenia (General disorders) | 3 (3)
Insomnia (General disorders) | 2 (3)
Rigors/chills (Nervous system disorders) | 3 (3)
Weight loss (Gastrointestinal disorders) | 13 (32)
Dermatology/skin/other (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (8)
Hair loss/alopecia scalp or body (Skin and subcutaneous tissue disorders) | 9 (12)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (3)
Rash/hand foot skin reaction (Skin and subcutaneous tissue disorders) | 4 (9)
Anorexia (Gastrointestinal disorders) | 22 (53)
Constipation (Gastrointestinal disorders) | 8 (10)
Dehydration (Gastrointestinal disorders) | 20 (36)
Diarrhea (Gastrointestinal disorders) | 18 (33)
Mucositis/stomatitis/oral cavity (Gastrointestinal disorders) | 13 (33)
Nausea (Gastrointestinal disorders) | 21 (67)
Taste alteration/dysgeusia (Gastrointestinal disorders) | 11 (16)
Vomiting (Gastrointestinal disorders) | 17 (39)
Hemorrhage/pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Albumin serum low/hypoalbulinemia (Metabolism and nutrition disorders) | 2 (2)
Alkaline phosphatase (Metabolism and nutrition disorders) | 4 (5)
ALT/SGPT/serum glutammic pyruvic transaminase (Metabolism and nutrition disorders) | 2 (3)
AST/SGOT/serum glutamic oxaloacetic transaminase (Metabolism and nutrition disorders) | 2 (3)
Calcium/serum low hypocalcemia (Metabolism and nutrition disorders) | 18 (30)
Glucose serum high hyperglycemia (Metabolism and nutrition disorders) | 4 (12)
Magnesium serum low hypomagnesemia (Metabolism and nutrition disorders) | 12 (21)
Potassium serum low/hypokalemia (Metabolism and nutrition disorders) | 6 (8)
Mood alteration/depression (Nervous system disorders) | 3 (3)
Neuropathyy sensory (Nervous system disorders) | 2 (2)
Pain/abdomen nonspecific (General disorders) | 12 (21)
Pain back (General disorders) | 2 (2)
Pain/head/headache (General disorders) | 2 (2)
Pain/throat/pharynx/larynx (General disorders) | 2 (2)
Pain/other (General disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes